CLINICAL TRIAL: NCT06089811
Title: A Nutritional Intervention to Prevent Stress Induced Intestinal Hyper-Permeability
Acronym: HYPERNUTRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Prof., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: S66915
Record Dates: First submitted 2023-10-10; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological | interventions — Prebiotics; Tryptophan

STUDY DESIGN:
Intervention Model Description: The present study is a parallel group randomized controlled trial (RCT) aiming to investigate whether two nutritional interventions (prebiotics and L-tryptophan) can improve intestinal barrier function, attenuate the stress response, affect cognitive processes, and prevent stress-induced hyperpermeability. Participants will perform 2 study visits of 3h each and with 28 days in between, in which participants will be subjected to the L-PAST. During the L-PAST, 3 cognitive tasks will be administered. Moreover, participants will be asked to take a basal intestinal permeability test at home 2 days before the test days.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, and personnel involved in data analyses are blinded to the intervention. Unblinding occurs after all data has been collected AND analysed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prebiotic (Experimental)
  Interventions: Dietary Supplement: Prebiotic
- L-Tryptophan (Experimental)
  Interventions: Dietary Supplement: L-Tryptophan
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Prebiotic — Group 1 (prebiotic and placebo L-tryptophan): prebiotic (oligofructose, Orafti®P95, 20g/day) and placebo L-tryptophan (microcrystalline cellulose, 3g/day)
  Arms: Prebiotic
Dietary Supplement: L-Tryptophan — Group 2 (placebo prebiotic and L-tryptophan): L-tryptophan (3g/day) and placebo prebiotic (microcrystalline cellulose, 20g/day)
  Arms: L-Tryptophan
Dietary Supplement: Placebo — Group 3 (placebo prebiotic and placebo L-tryptophan): placebo prebiotic (microcrystalline cellulose, 20g/day) and placebo L-tryptophan (microcrystalline cellulose, 3g/day).
  Arms: Placebo

SUMMARY:
The interaction between the gut microbiome, the intestinal barrier, and the host plays an important role in human health. The integrity of the intestinal barrier is essential to protect against translocation of food antigens and immunostimulatory microbial metabolites from the gut lumen. Accumulating studies show that stress may negatively affect the intestinal barrier function. In a previous study, the investigators developed the Leuven Prolonged Acute Stress Test (L-PAST), which combines physical (cold water), mental (arithmetic), and social (negative feedback) aspects of stress for a prolonged (2h) time. In the current study the investigators would like, as a first aim, to investigate whether the L-PAST 1) increases intestinal permeability compared to baseline intestinal permeability, and 2) whether a nutritional intervention can improve baseline intestinal permeability as well as intestinal permeability after exposure to the L-PAST in both healthy females and men. As a second aim of the present study, the investigators would like to investigate whether prebiotics and/or L-tryptophan can attenuate the cortisol response to stress. Lastly, as acute psychosocial stress impairs cognitive functions, the investigators would like as a third aim to investigate whether prebiotics and/or L-tryptophan supplementation may prevent these impairments.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 till 40 years (both included)
* BMI range: 18.5 - 25 kg/m²
* Females: Use of contraceptives, and have to use the current contraceptive method for at least 4 months. A regular menstrual cycle (between 25 and 35 days; if not using oral contraceptives)
* Subject is willing to not consume caffeine, or alcohol, to refrain from smoking, and not to engage in heavy physical exercise three days before the test days, as well as to not consume dairy products and chewing gum the day before and the day of the test days
* Subject is willing to not take any non-steroidal anti-inflammatory drugs (NSAIDs) two weeks before the test days (see Appendix G for an overview of NSAIDs)
* Subject, upon briefing of the content of the present study, fully understands and agrees to its objective and has given written (dated and signed) informed consent form to take part in the study
* Subject is able to communicate well with the investigator and follow instructions given by the investigator

Exclusion Criteria:

* Subject has a previous or current neurological, psychiatric, gastrointestinal, or endocrine disorder, or other relevant medical history
* Subject has one or more diagnoses based on the MINI international neuropsychiatric interview
* Subject has one or more diagnoses based on the ROME-IV for GI disorders
* Subject uses regular medication (i.e., anti-allergy medication, PPI's, and medication that can affect gut motility), currently or recently (in the last 2 weeks) (except for oral contraceptives)
* Subject has used recreational drugs in the past 6 months
* Subject consumes regularly (>1/week) more than 3 units of alcohol per day
* Subjects smokes >7 cigarettes per week
* Subject has to work in night-shifts
* Subject is pregnant or lactating
* Subject has previous experience with the stress test used in the study
* Subject has taken prebiotics or probiotics in the last month
* Subject has taken antibiotics in the last 3 months
* Subjects consumes >25g of fiber per day in their habitual diet

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Executive functions during a prolonged stress task (the Leuven Prolonged Stress Test) | Measured during the stress induction task during both the pre-intervention visit and immediately after the 4 week intervention.
  Working memory, cognitive flexibility, and response inhibition. Working memory will be assessed using the forward digit span. Cognitive flexibility will be assessed using the Wisconsin Card Sorting Test. Response inhibition will be assessed using the Stop Signal Task.

SECONDARY OUTCOMES:
Intestinal permeability after a prolonged stress task (the Leuven Prolonged Stress Test) | Measured at the pre-intervention and immediately after the 4 week intervention.
  Intestinal permeability will be measured using the lactulose-mannitol test. The lactulose-mannitol ratio will be calculated and used as a measure for small intestinal permeability. Fractional excretion of lactulose and mannitol will also be assessed.
Stress response to a prolonged stress test (the Leuven Prolonged Stress Test) | During the stress task (at multiple time points during 120 min), measured at the pre-intervention and immediately after the 4 week intervention.
  Cortisol, blood pressure, and subjective stress. Cortisol will be measured in saliva. Subjective stress will be measured using a Visual Analogue Scale (VAS)

OTHER OUTCOMES:
Intestinal permeability baseline | Measured 2 days before the pre-intervention and immediately after the 4 week intervention.
  Intestinal permeability will be measured using the lactulose-mannitol test. The lactulose-mannitol ratio will be calculated and used as a measure for small intestinal permeability. Fractional excretion of lactulose and mannitol will also be assessed.
Short chain fatty acids | Measured for 3h during the pre-intervention and immediately after the 4 week intervention.
  Short chain fatty acids will be measured both in feces and serum.
Tryptophan metabolites | Measured in blood for 3h during the pre-intervention and immediately after the 4 week intervention. Urine will be collected 3 days prior to the pre-intervention and immediately after the 4 week intervention.
  Tryptophan metabolites (kynurenine and indole pathway) will be measured in urine and blood.
Inflammatory cytokines | Measured at the pre-intervention and immediately after the 4 week intervention.
  Including interleukin (IL)-1β, IL-6, IL-10, IL-13, interferon (IFN)-γ, and tumor necrosis factor (TNF)-α
Subjective pain response to the prolonged stress test | Measured during the stress induction task during both the pre-intervention visit and immediately after the 4 week intervention.
  The subjective pain response to the prolonged stress task (Leuven Prolonged Stress Test) will be measured using a Visual Analogue Scale (VAS) (1-100)
Cognitive reactivity to failure response to the prolonged stress test | Measured during the stress induction task during both the pre-intervention visit and immediately after the 4 week intervention.
  Cognitive reactivity to failure response to the prolonged stress task (Leuven Prolonged Stress Test) will be assessed using two rating scales on a scale of 0 to 100. On one scale, 0 means 'I feel much less self-assured than before, 50 means 'I feel as self-assured as before, and 100 means 'I feel much more self-assured than before'. On the other scale, 0 means 'I think I'm not good at anything at all, 50 means 'I still think the same about myself', and 100 means 'I think I can achieve anything'.
Perceived Stress Scale (PSS) | Measured at the pre-intervention and immediately after the 4 week intervention.
  The Perceived Stress Scale (PSS) is a 14-item instrument designed to measure the degree to which situations in one's life are appraised as stressful. It provides a tool for examining issues about the role of appraised stress levels in the etiology of disease and behavioral disorders. The scale is designed such that it asks the respondent to rate the frequency of his/her feelings and thoughts related to events and situations that occurred over a selected time-frame. Notably, high PSS scores have been correlated with higher biomarkers of stress, such as cortisol.
Gastrointestinal symptom rating scale (GSRS) | Measured at the pre-intervention and immediately after the 4 week intervention.
  The Gastrointestinal Symptom Rating Scale (GSRS) is a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhea and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms. The reliability and validity of the GSRS are well-documented, and norm values for a general population are available.
Patient Health Questionnaire 9 (PHQ-9) | Measured at the pre-intervention and immediately after the 4 week intervention.
  The Patient Health Questionnaire - 9 (PHQ-9) is a 9-item questionnaire based on the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV). This self-report measure determines the severity of depression symptoms and is frequently used to monitor changes in symptom severity over time in non-psychiatric settings. Subjects are asked to rate each of the items on a scale of 0 to 3 on the basis of how much a symptom has bothered them over the last 2 weeks (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day).
Generalized Anxiety Questionnaire 7 (GAD-7) | Measured at the pre-intervention and immediately after the 4 week intervention.
  The Generalized Anxiety Questionnaire (GAD-7) is a 7-item questionnaire based on the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV). This self-report measure reflects the frequency of anxiety symptoms over the past 2 weeks. Subjects are asked to rate each of the items on a scale of 0 to 3 on the basis of how much a symptom has bothered them over the last 2 weeks (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day).

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven/ UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided